CLINICAL TRIAL: NCT05894954
Title: EVANTHEA TRIAL: a Pragmatic, Randomized, Controlled Trial to Evaluate the Effectiveness of a Precision Medicine Treatment Approach for Early Dementia and Mild Cognitive Impairment
Brief Title: Precision Medicine Approach for Early Dementia & Mild Cognitive Impairment
Acronym: EVANTHEA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alzheimer's Prevention and Reversal Project, Inc. (Other)
Collaborators: Four Winds Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EVANTHEA-2023
Record Dates: First submitted 2023-04-30; First posted 2023-06-08 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Mild Cognitive Impairment; Dementia, Mild
Keywords: Mild Cognitive Impairment; Early-stage dementia; Mild dementia; Alzheimers Disease; Short term memory; Mental recall; MCI; Word finding difficulty
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Lymphoma, Follicular; Alzheimer Disease; Anomia | interventions — Hormones; Standard of Care; Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two treatment groups. Group A is Precision Medicine Approach and Group B is the Standard-of-Care (Control) Group. Both groups will be on study for 9 months. Biomarker tests and cognition tests will be conducted in both groups at baseline, defined visits during the study and again at end of the 9-month period.
Who Masked: Outcomes Assessor
Masking Description: A masked psychometrician will conduct the Montreal Cognitive Assessments (MoCA) and Alzheimers Questionnaires.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Precision Medicine) (Experimental): Precision Medicine approach starts with a battery of tests and questionnaires to determine a person's underlying causes of cognition impairment. A custom treatment program is developed and prescribed by the investigator based on the test results and includes a combination of: supplements, medications, hormone therapy, dietary changes, exercise program, brain exercises, stress management, sleep tracking. Additional treatments may include QEEG and photobiomodulation, neurostimulation, neurofeedback and/or hyperbaric oxygen treatment (additional treatment are only available at select sites). Participants in this Group will also be supported in their program by a nutritionist, health coach, and fitness trainer, in addition to the study doctor. Tracking of study activities may also be required in the form of diaries, and devices will be used to track some of their activities such as sleep, stress, diet and exercise.
  Interventions: Dietary Supplement: Precision Medicine Approach; Combination Product: Hormones and Medications tailored to lab tests, combined with devices that support stress management and brain exercises; Behavioral: Lifestyle including diet, exercise, stress management
- Group B (Standard-of-Care) (Active Comparator): Standard-of-care treatment will be based on the practice guideline of hte Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology. Participants in this group will be guided according to the recommendations which include recommending:
  * participation in cognitively and socially-stimulation activities
  * regular exercise
  * ensuring quality sleep including treatment of any sleep apnea
  * control of any modifiable risk factors such as blood pressure, diabetes, cholesterol, and avoidance of tobacco use
  * evaluation by a primary care physician
  * adherence to a healthy and balanced diet
  * consult a neurologist or primary care physician regarding use of medications
  * consult with their primary care physician to identify any worsening conditions
  Interventions: Behavioral: Standard-of-Care

INTERVENTIONS:
Dietary Supplement: Precision Medicine Approach — Precisions Medicine Approach involves a combination of medicines, dietary supplements, lifestyle changes, and diagnostics
  Other Names: ReCODE
  Arms: Group A (Precision Medicine)
Combination Product: Hormones and Medications tailored to lab tests, combined with devices that support stress management and brain exercises — Tailored Medications and Devices to address imbalances per lab results, known to affect cognitive function:
  Potential Devices: Oura Ring, Continuous Glucose Monitor, Keto-Mojo, and Heartmath Inner Balance. Few may receive Hyperbaric Oxygen Treatment, neurostimulation, neurofeedback, neurostimulation to reduce stress and relax the body), photobiomodulation (light therapy), or CPAP.
  Atrophic subtype support may include: estradiol, progesterone, testosterone, DHEA, pregnenolone, levothyroxine, liothyronine, hydrocortisone.
  Bacterial or Viral infection treatment may include: Doxycycline, Minocycline, Nitazoxanide, Hydroxychloroquine, Rifampin, Dapsone, Azithromycin, Tetracycline, Benzathine Penicillin G, Methylene Blue, Nystatin, Clotrimazole, Metronidazole, Valacyclovir, Acyclovir, Famciclovir, Shingles Vaccine Vascular treatments may include: antihypertensives, Ubrelvy, aspirin, Eliquis
  Arms: Group A (Precision Medicine)
Behavioral: Standard-of-Care — Participate in cognitively stimulating and social activities, exercise, sleep, control risk factors, adhere to a health diet, consult physician if conditions worsen
  Other Names: Academy of Neurology practice guidelines
  Arms: Group B (Standard-of-Care)
Behavioral: Lifestyle including diet, exercise, stress management — Combining a tailored diet, exercise and stress management program supported by coaching specialists
  Arms: Group A (Precision Medicine)

SUMMARY:
The goal of this clinical trial is to compare a precision medicine approach to the standard-of-care for people with mild cognitive impairment or early-stage dementia. Precision medicine approach starts with the completion of many tests and then the study doctor uses the test results to carefully prepare a treatment plan that is best for the individual person to help treat many of the underlying causes of mild cognitive impairment or early-stage dementia.

The main question the study aims to answer is:

• Does the precision medicine approach improve memory (cognitive function) better than the current standard-of-care treatment in people with mild cognitive impairment or early-stage dementia during a 9-month treatment period? This is a randomized clinical trial which means that a group of people that meet the study requirements will be assigned at random or by chance (like toss of a coin) to receive either the precision medicine treatment or the current gold standard (standard-of-care). People assigned to the precision medicine group will receive precision medicine for 9-months while those assigned to the standard-of-care group will follow that approach for 9-months, followed by an opportunity to receive up to six months of precision medicine, if desired.

Participants will be asked to:

* Have their blood drawn for extensive lab testing and collect urine and stool samples as well
* Carefully follow instructions received from their study doctor and study team
* Make lifestyle changes as prescribed by the study doctor and study team based on your precision medicine program
* Take supplements and medications prescribed by the study doctor.
* Once officially in the study (after meeting study entry or screening requirements), participate in ten (10) monthly visits with the study doctor, and other members of the study team as scheduled.
* Complete cognitive tests at scheduled visits during the study
* Have a study partner with you during visits and to help support you on the program Researchers will compare test results between the two study groups to see if the precision medicine approach improves those tests results over the time of the study, resulting in the improvement of cognition over a 9-month treatment period.

DETAILED DESCRIPTION:
The precision medicine treatment approach to be evaluated in this clinical trial is a novel, functional, lifestyle intervention for the treatment of mild cognitive impairment or early-stage dementia. The protocol focuses on optimization of a diverse set of metabolic parameters coupled with lifestyle medicine and clinical nutrition strategies that address the mismatch in these contributors. The approach is personalized for each participant and based on more than 150 data points, including lab evaluations, brain scans, genomic evaluation, cognitive testing, and a detailed medical and family history. Importantly, this progressive treatment approach is based on continued optimization through iterative treatment and metabolic characterization.

The precision medicine treatment approach includes a core set of interventions (Precision Medicine-Core) and a set of interventions that are based on the clinical subtype of dementia (Precision Medicine-Cognitive Subtypes). All participants randomized to the precision medicine treatment approach group will receive the core treatment program. The elements of the core treatment program include diet, physical exercise, mental exercise, sleep optimization, and stress reduction.

In addition, all participants randomized to the precision medicine treatment approach will be evaluated for all putative or potential underlying drivers of dementia including: 1) inflammatory factors (Type 1 Inflammatory), 2) glycotoxic factors (Type 1.5 Glycotoxic), 3) atrophic factors (Type 2 Atrophic), toxic factors (Type 3 Toxic), vascular factors (Type 4 Vascular), and traumatic factors (Type 5 Head Trauma).

This study will use a pragmatic, randomized, multicenter, control group design in which participants will be randomized to a 9-month precision medicine treatment approach or a 9-month standard-of-care treatment approach. Participants in the standard-of-care group will receive the standard-of-care mild cognitive impairment and early-stage dementia. Following completion of the 9-month intervention period, participants in the standard-of-care group will be eligible to receive the precision medicine treatment approach.

During the course of the 9-month precision medicine treatment approach, participants and study partners will be scheduled for regular visits with members of the study team at each practice. These visits will be scheduled at approximately 4-week intervals following randomization. Cognitive function tests will be performed at baseline (Visit 1), Month 3 (Visit 4), Month 6 (Visit 7), and Month 9 (Visit 10). Cognitive testing includes the MoCA to be performed by a blinded psychometrician prior to randomization and then 1-2 weeks before the 3-, 6-, and 9-month visits. The CNS Vital Signs will be performed by each staff at each of the six participating sites. Participants in the standard-of-care treatment group will complete a similar set of visits at the same intervals during this time.

A final follow-up visit will occur within 4 weeks of completion of Visit 10 to complete all effectiveness and safety follow-up assessments. Following completion of the final follow-up visit, all participants in the standard-of-care treatment group will be eligible for initiation of a 6-month precision medicine treatment approach. Safety data will be collected for participants in both groups through completion of the 6-month precision medicine intervention period for participants initially randomized to the standard-of-care treatment group. Periodic unblinded safety reviews are planned at approximately 1-month intervals for the full duration of the trial. These reviews will be conducted by the Study Oversight and Safety Review Committee.

Participants will be enrolled from six geographically-diverse clinical practices and randomized to either the precision medicine treatment approach (Group A) or the standard-of-care control group (Group B). The population to be enrolled will be heterogenous in terms of demographic and clinical characteristics of their cognitive dysfunctions. In addition, the precision medicine intervention will be heterogenous because, by definition, precision medicine is personalized to target the specific metabolic abnormalities that are identified in each participant as uniquely associated with mild cognitive impairment or early-stage dementia. Given the real-world settings, heterogeneity in study participants, and heterogeneity of the specific precision medicine components, a pragmatic, randomized, controlled trial will provide the best evaluation of the precision medicine treatment approach while offering maximum external validity and the ability to generalize findings from this study to precision medicine practice settings and patients who are treated in the US.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed informed consent
* Adults of any gender, race, or ethnicity and aged 45 to 76 years at time of enrollment
* Cognitive impairment or early-stage dementia as demonstrated by combination of AQ-21 score >4 and either:
* MoCA 18-26, inclusive, or
* greater than or equal 2 scores in the bottom 50th percentilve for NCI or Executive Function, Verbal, Visual, or Composite sub-tests
* Proficient in spoken and written English for informed consent and study procedures
* Have a willing and able study partner to support participant with compliance and all aspects of teh protocol and provide input for subjective ratings of the participant's cognitive status. The study partner must interact with teh participant frequently (live with or have daily contact with participant), and have sufficiently close relationship to observe and understand participant's difficulties with memor and activities of daily living.
* All exisiting medical conditions and any current medication dosages must be stable
* Have regular access to computer and internet connection and an iOS or Android Smartphone or tablet capable of connecting to devices and applications used in the study
* Ability to use a computer and web interface, or have readily available assistance to facilitate the use of a computer and web interface
* Ability to converse with a coach or provider virtually to access the virtual coaching aspects of the treatment approach
* Willing and able to follow the protocol procesured and testing, including changes in diet, lifestyle, supplements, and medications
* Willing to have at least one home visit by the study health coach, including home evaluation for toxins or mold
* Willingness to remediate and/or move away from identifies sources of toxicity such as molds or other toxins or infections or dental decay
* Willingness to comply with COVID prevention precautions
* Participants taking Aricept will be considered if they have been using Aricept for at least 90 days prior to study adminission. Must be on a stable dose for at least 90-days prior to screening and agree to remian on the same dose throughout the course of the study.
* Women who are premenopausal and sexually active must be willing to use appropriate contraception and have repeated pregnancy tests as indicated
* Willing to have an MRI and coronary artery calcium scan
* Live within 1-1.5 hours of the study site
* Women only: willing to complete the health screening exams and remediate any health issues detected during these screening exams: 1) Mammogram within 12 months of randomization; 2) Pelvic exam within 12 moths for women less than 60 years or pelvic exam within 24 months if 60 years or older.

Exclusion Criteria:

* Presence of any uncontrolled major medical illness, seizures, or cardiovascular disease
* Diagnosis of Type 1 Diabetes
* Presence of any major psychiatric diagnoses that impact the performance of activities of daily living or functioning, other than those related to cognitive decline
* Use of psychoactive medications known to impact cognition, unless willing and eligible to discontinue
* Use of chronic anticoagulation therapy, other than prophylactic aspirin or proteolytic enzymes, or a history of recurrent deep vein thrombosis
* MRI findings of hydrocephalus, focal stroke, extinsive white matter disease or brain tumor
* Prior traumatic brain injury of sufficient severity to impact functioning on a regular basis
* Diagnosis of cancer in past 5 years, or any history or breast cancer; exclusive of melanoma skin cancers or ductal carcinoma in situ.
* Positive test for HIV, Hepatitis C, or RPR (rapid plasma reagin)
* Menopausal and perimenopausal women who are unwilling or unable to use bioidentical hormone replacement therapy
* Positive preganance test
* Presence of an existing daignosis of non-Alzheimer's neurodegenerative disorders such as Lewy Body Disease, Frontotemporal Disease, Chronic Traumatic Encephalopathy, Korsakoff's Syndrome, etc.
* A diagnosis of cerebrovascular disease as the primary cause of cognitive impairment or early-stage dementia
* Lack of adequate support from a study partner to assist with study adherence
* Inability to exercise
* Inabilty to use a computer with or without assistance; or no computer access
* Plans to travel or be away from home for more than 2 weeks during the course of the 9-month study
* Previous treatment using dietary changes, comprehensive nutritional support, ReCODE Program, or similar methodology such as functional, integrative, or systems medicine at a level considered by the investigator to interfere with the study goals
* Any contraindication to enclosed MRI
* Unwilling or unable to comply with general study procedures
* Current user of tobacco
* Unwilling or unable to remediate or move away from identified sources of toxicities (molds, toxins, infections, dental decay)
* Use of Aricept off-label
* Two or more CNS-Vital Sign tests are invalid at baseline

Ages: 45 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Changes in mean Montreal Cognition Assessment (MoCA) scores over 9 months | Baseline and Months 3, 6, and 9 (end of study treatment)
  Compare changes over time between Group A and Group B in mean MoCA scores over 9 month treatment period
Changes in mean CNS Vital Signs Neurocognitive Index Scores over 9 months | Baseline and Months 3, 6, and 9 (end of study treatment)
  Compare changes over time in mean score on the CNS Vital Signs Neurocognitive Index over 9 month treatment period. Standard scores are used. 100 is the mean score with standard deviation of 15. No min/max value for the Index. Standard scores are normal distribution but there is a limit to human performance, towards 200. Higher score over time is better outcome.

SECONDARY OUTCOMES:
Changes over time in mean score on the Alzheimer's Questionnaire-21 (AQ-21) / Alzheimer's Questionnaire-20 (AQ-20) | Baseline and Months 3, 6, and 9 (end of study treatment)
  Compare changes over time between Group A and Group B in mean Alzheimer's Questionnaire scores. AQ-21 is baseline; AQ-20 is a modified version of the AQ-21 to address changes from baseline. The AQ© total score is based on the sum of points for items with a yes response. The range of possible scores is 0 to 27. Score interpretation: A score of four points or less is regarded as normal. A score between five and 14 points inclusive suggests mild cognitive impairment. A score of 15 or more points suggests dementia. Lower score over time is a better outcome.
Changes over time in mean score on the Patient-reported Outcome Measurement Information System (PROMIS-10). | Baseline and Month 9 (end of study treatment)
  Evaluate Group A treatment compared with Group B treatment with regard to changes over time in mean PROMIS-10 score. The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. The possible score ranges from 0 to 20 points in each case. 0 points represent the patient's most severe physical and/or mental impairment, while 20 points represent the best possible state of health.
Discontinuation rates | Throughout 9-month study treatment period
  Evaluate acceptability of the precision medicine intervention approach by comparing discontinuation rates in Group A and Group B participants
Safety: Type, frequency, severity, relatedness, and expectedness of adverse events and serious adverse events. | Throughout 9-month study treatment period
  Determine the safety of the Group A treatment compared with Group B treatment based on the type, frequency, severity, relatedness, and expectedness of adverse events and serious adverse events.

OTHER OUTCOMES:
Changes over time in findings on volumetric magnetic resonance imaging (MRI). | Baseline and Month 9 (end of study treatment)
  Compare the impact of a Group A treatment approach with Group B treatment in regards to changes over time in findings on volumetric magnetic resonance imaging (MRI).
Change in serum biomarker, methylation epigenetics. | Baseline and Month 9 (end of study treatment)
  Compare changes in methylation epigenetic results between Group A and Group B participants at the same timepoints, beginning and end of treatment.
Changes in serum biomarker, P-tau. | Baseline and Month 9 (end of study treatment)
  Compare changes P-tau results between Group A and Group B participants at the same timepoints, beginning and end of treatment. Lowering of P-Tau over course of the study is positive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dale Bredesen, MD, Study Chair — Alzheimer's Prevention and Reversal Project, Inc.; Kat Toups, MD, Principal Investigator — Bay Area Wellness
Locations (6):
- United States (6):
  - True Health Center for Functional Medicine, Folsom, California
  - Ann Hathaway, MD, San Rafael, California
  - Bay Area Wellness, Walnut Creek, California
  - Rezilir Health, Hollywood, Florida
  - Kemper Cognitive Wellness, Rocky River, Ohio
  - MaxWell Clinic, PLC, Brentwood, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toups K, Hathaway A, Gordon D, Chung H, Raji C, Boyd A, Hill BD, Hausman-Cohen S, Attarha M, Chwa WJ, Jarrett M, Bredesen DE. Precision Medicine Approach to Alzheimer's Disease: Successful Pilot Project. J Alzheimers Dis. 2022;88(4):1411-1421. doi: 10.3233/JAD-215707. PMID 35811518
- [Background] Bredesen DE, Amos EC, Canick J, Ackerley M, Raji C, Fiala M, Ahdidan J. Reversal of cognitive decline in Alzheimer's disease. Aging (Albany NY). 2016 Jun;8(6):1250-8. doi: 10.18632/aging.100981. PMID 27294343
- [Background] Rao RV, Kumar S, Gregory J, Coward C, Okada S, Lipa W, Kelly L, Bredesen DE. ReCODE: A Personalized, Targeted, Multi-Factorial Therapeutic Program for Reversal of Cognitive Decline. Biomedicines. 2021 Sep 29;9(10):1348. doi: 10.3390/biomedicines9101348. PMID 34680464
- [Background] Bredesen DE. Reversal of cognitive decline: a novel therapeutic program. Aging (Albany NY). 2014 Sep;6(9):707-17. doi: 10.18632/aging.100690. PMID 25324467
- [Background] McMaster M, Kim S, Clare L, Torres SJ, D'Este C, Anstey KJ. Body, Brain, Life for Cognitive Decline (BBL-CD): protocol for a multidomain dementia risk reduction randomized controlled trial for subjective cognitive decline and mild cognitive impairment. Clin Interv Aging. 2018 Nov 21;13:2397-2406. doi: 10.2147/CIA.S182046. eCollection 2018. PMID 30538436
- [Background] Ross MK, Raji C, Lokken KL, Bredesen DE, Roach JC, Funk CC, Price N, Rappaport N, Hood L, Heath JR. Case Study: A Precision Medicine Approach to Multifactorial Dementia and Alzheimer's Disease. J Alzheimers Dis Parkinsonism. 2021;11(Suppl 5):018. Epub 2021 Aug 25. PMID 35237464
- [Background] Shetty P, Youngberg W. Clinical Lifestyle Medicine Strategies for Preventing and Reversing Memory Loss in Alzheimer's. Am J Lifestyle Med. 2018 May 11;12(5):391-395. doi: 10.1177/1559827618766468. eCollection 2018 Sep-Oct. PMID 30283265
- See also: Published book describing basis for the precision medicine approach used in this trial — http://www.penguinrandomhouse.com/books/551532/the-end-of-alzheimers-by-dale-e-bredesen-md/